CLINICAL TRIAL: NCT01362257
Title: An Open-label, Two Period Study to Determine the Excretion Balance and Pharmacokinetics of 14C-GSK573719, Administered as Single Dose of an Oral Solution and an Intravenous Infusion, to Healthy Male Adults
Brief Title: A Study to Determine the Excretion Balance and Pharmacokinetics of 14C-GSK573719
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 112014
Record Dates: First submitted 2011-05-26; First posted 2011-05-30 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 14C-GSK573719 Oral Solution (Experimental): single dose of 1000µg
  Interventions: Drug: Treatment Period 2 - Oral dose of GSK573719
- 14C-GSK573719 IV Solution (Experimental): single dose of 65µg
  Interventions: Drug: Treatment Period 1 - IV dose of GSK573719

INTERVENTIONS:
Drug: Treatment Period 1 - IV dose of GSK573719 — single dose of 65µg
  Arms: 14C-GSK573719 IV Solution
Drug: Treatment Period 2 - Oral dose of GSK573719 — single dose of 1000µg
  Arms: 14C-GSK573719 Oral Solution

SUMMARY:
This will be a two-period, open-label study conducted at a single site. Six healthy male subjects will participate in the study to ensure at least four fully evaluable subjects. Each subject will receive a single 1000 μg (microgram) oral dose containing 50 μCi (Micro Curie) of [14C]-GSK573719 and a 65 μg intravenous infusion containing 7.1 μCi of [14C]-GSK573719. Whilst subjects are in-house, urine and faecal samples will be collected for a minimum of 168 hours (7 days) after dosing or for up to 240 hours (10 days) depending on the amounts of radioactivity still being excreted after Day 5. Faecal sample collection may continue at home for up to 14 days. Bile samples will be collected using Entero-Test string sampling of duodenal bile. Whole blood and plasma samples will be collected at various sample times after dosing to measure parent drug (plasma only) and total radiolabelled drug related material (blood and plasma). Urine and faeces aliquots will be taken to measure total radiolabelled drug-related material. Samples of urine, faeces and plasma will be transferred into a separate study to characterize and, where possible, quantify metabolites in these matrices.

DETAILED DESCRIPTION:
This will be a single-centre, open-label, two period study in healthy male subjects. Each subject will participate in two separate dosing periods. In the first dosing period, each subject will receive a 65 μg single dose of intravenous infusion containing 7.1 μCi of [14C]-GSK573719 administered over 30 minutes. In the second dosing period, each subject will receive a single 1000 μg oral dose containing 50 μCi of [14C]-GSK573719. Each study period will involve an admission to the CRO (clinical research organisation) unit of between 7 and 10 days. The two dosing periods will be separated by a wash-out of at least 28 days between doses. Screening will occur within 30 days prior to the first dosing period. Each subject will be admitted to the clinical unit on the afternoon of Day -1. Whilst subjects are in-house, blood, urine and faecal samples will be collected for a minimum of 168 hours (7 days) after dosing or for up to 240 hours (10 days), depending on amounts of radioactivity still being excreted after day 5. Liquid scintillation counts (LSC) will be performed daily on the 24-hour urine pools and 24-hour faeces homogenates after Day 5 to measure total radioactivity concentrations. If less than 1% of the dose is excreted in each 24 hour period on Day 6 and Day 7 for a given subject, that subject will be discharged on Day 8, after the results of the LSC counts are available, and no further samples will be collected. If excretion is higher than 1%, or if the results are inconclusive, the subject will remain in-house, and urine and faecal collections will continue at 24 hour intervals, until excretion is less than 1% on Day 8, 9 or 10; again subjects will be discharged after the results of the LSC counts are available. On the morning of Day 11, all remaining subjects will be discharged from the clinic and subjects will be notified by phone as to whether they need to continue faecal collection at home. In the event that excretion is still higher than 1% upon discharge on Day 11, subjects will continue to collect faecal samples only, at home, at 24 hour intervals up to and including Day 14. Samples collected at home will be returned to the clinic every 2-3 days. The Entero-Test will be used in Treatment Period 1 only (IV dosing). The Entero-Test will be inserted at approximately 3.5 hours pre-dose while subjects are in a fasted state and removed at approximately 2.5 hours post-dose on day 1. At approximately 0.5 hours post-dose (i.e. two hours prior to string withdrawal) a food cue will be used to stimulate gall bladder emptying. Safety data collected will include spontaneous AE (adverse event) reporting, 12-lead ECG (electrocardiogram), vital signs, nursing/physician observation and safety laboratory tests. Subjects will complete follow up assessments within 8-12 days of their last dose (this may happen on the day of discharge from the unit). Final follow up contact will then be via telephone call to the subjects 2 to 3 days after final sample collection. The duration of the study will be approximately 11 to 12 weeks for each subject.

ELIGIBILITY:
Inclusion:

AST (Aspartate aminotransferase), ALT (Alanine aminotransferase), alkaline phosphatase and bilirubin ≤ 1.5xULN (Upper limit of normal) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%) Healthy, non-smoking male subjects, 30-55 years old inclusive Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in Section 8.1 Body Mass Index (BMI) within the range 18.5-29.0 kg/m2 (inclusive) Capable of giving written informed consent Average QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block Available to complete the study A history of regular bowel movements

Exclusion:

A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening A positive test for HIV (Human Immunodeficiency Virus) antibody Current or chronic history of liver disease, or known hepatic or biliary abnormalities Any clinically relevant abnormality identified on the screening medical assessment laboratory examination or 12-lead ECG (Electrocardiogram) Subjects with a positive urine test for drugs of abuse or alcohol at screening or prior to study medication administration Positive urine cotinine at screening History of regular alcohol consumption within 6 months of the study Treatment with an investigational drug within 60 days or 5 half-lives preceding the first dose of study medication Subjects who have had exposure to more than four new chemical entities within 12 months prior to the first dosing period Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 7 days or 5 half-lives prior to the first dose of study medication Subjects who have received prescription medication within 14 days prior to the first dose of study drug. Subjects may still be entered into the study, if the prescription medication will not interfere with study procedures or compromise safety Donation of blood in excess of 500mL within 56 days prior to the first dose of study medication Participation in a clinical trial involving administration of 14C-labelled compound(s) within the last 12 months Subjects who have received a total body radiation dose of greater than 5.0 mSv or exposure to significant radiation in the 12 months prior to this study Previous history of active gastric or duodenal ulcer within 6 months prior to the first dose of study medication Any history of bleeding diathesis A pre-existing condition(s) interfering with normal gastrointestinal (GI) anatomy or motility or other GI dysfunction which may interfere with the absorption, distribution, metabolism or elimination of the study drug Surgical procedures on digestive tract An occupation which requires monitoring for radiation exposure, nuclear medicine procedures or excessive x-rays within the past 12 months History of anaphylaxis or anaphylactoid reactions, severe allergic responses to drugs History of sensitivity to any of the study medications Unwillingness or inability to follow the procedures outlined in the protocol Subject is mentally or legally incapacitated

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-04-29 (Actual); Primary Completion 2011-06-22 (Actual); Study Completion 2011-06-22 (Actual)

PRIMARY OUTCOMES:
AUC(0-∞), AUC(0-t), Cmax, tmax, λz and t1/2 of total drug-related material (radioactivity) and GSK573719 in plasma following intravenous and oral dosing | up to 8 days post-dose
  AUC(0-∞) = area under concentration time curve from time zero extrapolated to infinite time. AUC(0-t) = Area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration within a subject across all treatments. Cmax = Maximum observed concentration. tmax = Time of occurrence of Cmax. λz = Terminal phase rate constant. t1/2 = Terminal phase half life.
Urinary and faecal cumulative excretion as a percentage of the total radioactive dose administered over time | up to 14 days post dose

SECONDARY OUTCOMES:
Oral F (absolute bioavailability) | up to 8 days post dose
AUClast for oral dose, volume and clearance for intravenous dose | up to 8 days post dose
  AUC = Area under concentration-time curve
Characterisation and quantification of metabolites in plasma, urine, duodenal bile and faecal homogenates to be documented and performed by DMPK, GSK and the results will be reported in a separate report | up to 14 days post dose
Blood: plasma ratio of total drug related material (radioactivity) | up to 8 days post dose
Spontaneous AE reporting, 12-lead ECG, vital signs and safety laboratory tests | up to 14 days post dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Zuidlaren, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 112014 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/112014?search=study&search_terms=112014#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 112014 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112014 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112014 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112014 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112014 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112014 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112014 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register